CLINICAL TRIAL: NCT04307043
Title: Prospective Study on Geometric Parameters and Hemodynamic Reference Range of Neonatal Heart.
Brief Title: Study on the Geometric Parameters and Hemodynamic Reference Range of Neonatal Heart.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dan Fang Lu, Attending physician, Peking University Third Hospital
Other Study IDs: bysypediatric2020-1
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Echocardiography of Newborns
Keywords: Echocardiography, Heart, Neonatal, Reference range

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postnatal age
- General information and echocardiographic data: General information:(1)Record the gestational age, birth weight, length, delivery way, Apgar score, maternal pregnancy status, prenatal bleeding or not after admission.(2)PS use, ventilator mode, other illness and complications should be recorded during hospitalization. (3) Record the baby's heart rate, respiratory rate, blood pressure, body surface area on every check.

SUMMARY:
Perform bedside echocardiography on neonates (term and preterm infants) who were admitted to our neonatal department within 24 hours of birth, and establish a geometric reference range of neonatal cardiac ultrasound and explore the hemodynamic changes of early newborns.

Bedside echocardiography were performed to measure the diameter of each heart cavity and large vessels, velocity of each valve and aorta, wall thickness, left ventricular systolic function, right heart Tei index, Tricuspid Annular Plane Systolic Excursion(TPASE) of term and preterm infants respectively on 0 day, 3d, 7d of life and postmenstrual age of 30 weeks, 32 weeks, 34 weeks and 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Infants with normal hearts (infants with small patent fora-men oval or small patent ductus arteriosus were not excluded).

  2.Healthy preterm infant with no evidence of sepsis, renal failure. 3. Absence of other major congenital anomalies or syndromes 4. Prior written consent was obtained from the parents.

Exclusion Criteria:

* Infants with severe congenital malformations, either cardiac or non-cardiac.

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Babies born in the obstetrics department of Peking University Third Hospital and admitted to the neonatal ward.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Reference range of cardiac geometric parameters of preterm infants based on different gestational ages, weights, days of age and body surface area. | 0 day of life to PMA 36 weeks
Hemodynamic changes in full-term and preterm infants on 0~7days of life. | 0~7days of life

SECONDARY OUTCOMES:
Reference range of cardiac geometric parameters of full-term infants based on different weights, days of age and body surface area. | 0~7days of life

CONTACTS AND LOCATIONS:
Overall Officials: Yunfeng Liu, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jain A, El-Khuffash AF, Kuipers BCW, Mohamed A, Connelly KA, McNamara PJ, Jankov RP, Mertens L. Left Ventricular Function in Healthy Term Neonates During the Transitional Period. J Pediatr. 2017 Mar;182:197-203.e2. doi: 10.1016/j.jpeds.2016.11.003. Epub 2016 Nov 28. PMID 27908646
- [Background] Abushaban L, Vel MT, Rathinasamy J, Sharma PN. Normal Reference Ranges for Cardiac Valve Annulus in Preterm Infants. Pediatr Cardiol. 2016 Jan;37(1):112-9. doi: 10.1007/s00246-015-1247-9. Epub 2015 Sep 1. PMID 26321355
- [Background] Abushaban L, Vel MT, Rathinasamy J, Sharma PN. Normal Reference Ranges for Pulmonary Artery Diameters in Preterm Infants. Pediatr Cardiol. 2017 Oct;38(7):1377-1384. doi: 10.1007/s00246-017-1673-y. Epub 2017 Jul 7. PMID 28687889
- [Background] Abushaban L, Mariappa TV, Rathinasamy J, Sharma PN. Normal reference ranges for aortic diameters in preterm infants. J Saudi Heart Assoc. 2018 Apr;30(2):86-94. doi: 10.1016/j.jsha.2017.09.003. Epub 2017 Oct 1. PMID 29910578
- [Result] Levy PT, Dioneda B, Holland MR, Sekarski TJ, Lee CK, Mathur A, Cade WT, Cahill AG, Hamvas A, Singh GK. Right ventricular function in preterm and term neonates: reference values for right ventricle areas and fractional area of change. J Am Soc Echocardiogr. 2015 May;28(5):559-69. doi: 10.1016/j.echo.2015.01.024. Epub 2015 Mar 7. PMID 25753503